CLINICAL TRIAL: NCT07356011
Title: Improving Mediolateral Walking Balance With an Assistive Exoskeleton
Brief Title: Exoskeleton for Balance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jesse Dean, Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00135871; REGE22000170 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2025-12-08; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: walking; balance; exoskeleton
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: All participants will experience the same series of experimental sessions. Within individual sessions, the order in which different exoskeleton conditions are tested will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- xoskeleton Assistance Conditions (No Exoskeleton, Zero, Low, Medium, High Impedance) (Experimental): Participants in this arm will walk on a treadmill under several conditions. In one condition, they will not wear the exoskeleton. In other conditions, the exoskeleton will be set to zero, low, medium, or high impedance.
  Interventions: Device: No Exoskeleton; Device: Exoskeleton (zero impedance); Device: Exoskeleton (low impedance); Device: Exoskeleton (medium impedance); Device: Exoskeleton (high impedance)

INTERVENTIONS:
Device: No Exoskeleton — The participant will not wear an exoskeleton
Device: Exoskeleton (zero impedance) — The participant will wear an exoskeleton with zero impedance
Device: Exoskeleton (low impedance) — The participant will wear an exoskeleton with low joint impedance
Device: Exoskeleton (medium impedance) — The participant will wear an exoskeleton with medium joint impedance
Device: Exoskeleton (high impedance) — The participant will wear an exoskeleton with high impedance

SUMMARY:
Many people who have experienced a stroke have deficits in their walking balance. The long-term goal of this research is to develop an exoskeleton that can effectively improve walking balance, thus improving functional mobility.

DETAILED DESCRIPTION:
Walking balance is an important component of functional mobility, with post-stroke balance deficits contributing to a fall rate more than double that of age-matched controls. Unfortunately, traditional therapy approaches have not succeeded in addressing balance deficits or reducing fall risk, motivating the use of technology to fill this gap. Although assistive exoskeletons are a promising approach to improve post-stroke mobility, they have generally not been designed to control walking balance and agility. This limitation is a particular concern in the development of devices for people with stroke, as applying forces to "assist" some aspect of walking (including balance) can have unexpected negative effects. The project goal is to investigate the potential of exoskeleton assistance to improve walking balance that will be accepted by people with stroke. To this end, investigators will use a previously developed hip exoskeleton to quantify the effects of assisting gait stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a stroke at least 6 months prior to participation
* Evidence of dysfunction of the paretic lower limb (Fugl-Meyer lower extremity motor score < 34)
* At least 21 years of age
* Self-reported experience of a fall in the previous year, and/or a fear of falling
* Gait speed of at least 0.2 m/s
* Ability to walk on a treadmill without a cane or walker
* Ability to follow three step commands and communicate with experimenters to answer questions (e.g., regarding their balance confidence)
* Provision of informed consent

Exclusion Criteria:

* Resting blood pressure higher than 220/110 mm Hg
* History of unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living
* Preexisting neurological orders or dementia
* Legal blindness or severe visual impairment
* Presence of neglect
* History of DVT or pulmonary embolism within 6 months
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* Orthopedic injuries or conditions (e.g., joint replacements) in the lower extremities with the potential to alter the gait pattern

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Partial correlation (rSW) between mediolateral pelvis displacement and step width during unperturbed walking | Visit 2, anticipated average 1 week
  Mediolateral pelvis displacement will be quantified at the start of each step, and step width will be calculated at the end of each step. Across all steps, the partial correlation between these two metrics will be calculated - accounting for the mediolateral pelvis velocity. This will be done for steps taken with each leg independently.
Partial correlation (rSW) between mediolateral pelvis displacement and step width during speed perturbations | Visit 4, anticipated average 1 year
  Mediolateral pelvis displacement will be quantified at the start of each step, and step width will be calculated at the end of each step. Across all steps, the partial correlation between these two metrics will be calculated - accounting for the mediolateral pelvis velocity. This will be done for steps taken with each leg independently.
Partial correlation (rSW) between mediolateral pelvis displacement and step width during vision perturbations | Visit 4, anticipated average 1 year
  Mediolateral pelvis displacement will be quantified at the start of each step, and step width will be calculated at the end of each step. Across all steps, the partial correlation between these two metrics will be calculated - accounting for the mediolateral pelvis velocity. This will be done for steps taken with each leg independently.
Partial correlation (rSW) between mediolateral pelvis displacement and step width during mediolateral pull perturbations | Visit 4, anticipated average 1 year
  Mediolateral pelvis displacement will be quantified at the start of each step, and step width will be calculated at the end of each step. Across all steps, the partial correlation between these two metrics will be calculated - accounting for the mediolateral pelvis velocity. This will be done for steps taken with each leg independently.

SECONDARY OUTCOMES:
Partial correlation between mediolateral pelvis displacement and mediolateral foot placement (unperturbed walking) | Visit 2, anticipated average 1 week
  Mediolateral pelvis displacement will be quantified at the start of each step, and mediolateral foot placement relative to the pelvis will be calculated at the end of each step. Across all steps, the partial correlation between these two metrics will be calculated - accounting for the mediolateral pelvis velocity. This will be done for steps taken with each leg independently.
Average gluteus medius activity during stance phase (surface EMG) in unperturbed walking | Visit 2, anticipated average 1 week
  Average gluteus medius EMG activity will be calculated during the stance phase of walking. This will be calculated for each leg independently.
Average gluteus medius activity during swing phase (surface EMG) in unperturbed walking | Visit 2, anticipated average 1 week
  Average gluteus medius EMG activity will be calculated during the swing phase of walking. This will be calculated for each leg independently.
Rating of Perceived Stability (RPS) during unperturbed walking | Visit 2, anticipated average 1 week
  This patient reported outcome measure uses a validated scale for participants to self-report their perceived balance while walking.
Partial correlation between mediolateral pelvis displacement and mediolateral foot placement during speed perturbations | Visit 4, anticipated average 1 year
  Mediolateral pelvis displacement will be quantified at the start of each step, and mediolateral foot placement relative to the pelvis will be calculated at the end of each step. Across all steps, the partial correlation between these two metrics will be calculated - accounting for the mediolateral pelvis velocity. This will be done for steps taken with each leg independently.
Average gluteus medius activity during stance phase (surface EMG) with speed perturbations | Visit 4, anticipated average 1 year
  Average gluteus medius EMG activity will be calculated during the stance phase of walking. This will be calculated for each leg independently.
Average gluteus medius activity during swing phase (surface EMG) with speed perturbations | Visit 4, anticipated average 1 year
  Average gluteus medius EMG activity will be calculated during the swing phase of walking. This will be calculated for each leg independently.
Rating of Perceived Stability (RPS) with speed perturbations | Visit 4, anticipated average 1 year
  This patient reported outcome measure uses a validated scale for participants to self-report their perceived balance while walking.
Partial correlation between mediolateral pelvis displacement and mediolateral foot placement during vision perturbations | Visit 4, anticipated average 1 year
  Mediolateral pelvis displacement will be quantified at the start of each step, and mediolateral foot placement relative to the pelvis will be calculated at the end of each step. Across all steps, the partial correlation between these two metrics will be calculated - accounting for the mediolateral pelvis velocity. This will be done for steps taken with each leg independently.
Average gluteus medius activity during stance phase (surface EMG) with vision perturbations | Visit 4, anticipated average 1 year
  Average gluteus medius EMG activity will be calculated during the stance phase of walking. This will be calculated for each leg independently.
Average gluteus medius activity during swing phase (surface EMG) with vision perturbations | Visit 4, anticipated average 1 year
  Average gluteus medius EMG activity will be calculated during the swing phase of walking. This will be calculated for each leg independently.
Rating of Perceived Stability (RPS) with vision perturbations | Visit 4, anticipated average 1 year
  This patient reported outcome measure uses a validated scale for participants to self-report their perceived balance while walking.
Partial correlation between mediolateral pelvis displacement and mediolateral foot placement during mediolateral pull perturbations | Visit 4, anticipated average 1 year
  Mediolateral pelvis displacement will be quantified at the start of each step, and mediolateral foot placement relative to the pelvis will be calculated at the end of each step. Across all steps, the partial correlation between these two metrics will be calculated - accounting for the mediolateral pelvis velocity. This will be done for steps taken with each leg independently.
Average gluteus medius activity during stance phase (surface EMG) with mediolateral pull perturbations | Visit 4, anticipated average 1 year
  Average gluteus medius EMG activity will be calculated during the stance phase of walking. This will be calculated for each leg independently.
Average gluteus medius activity during swing phase (surface EMG) with mediolateral pull perturbations | Visit 4, anticipated average 1 year
  Average gluteus medius EMG activity will be calculated during the swing phase of walking. This will be calculated for each leg independently.
Rating of Perceived Stability (RPS) with mediolateral pull perturbations | Visit 4, anticipated average 1 year
  This patient reported outcome measure uses a validated scale for participants to self-report their perceived balance while walking.
Change in mediolateral foot placement (cm) during pull perturbations relative to unperturbed steps | Visit 4, anticipated average 1 year
  The change in mediolateral foot placement locations between steps with and without pull perturbations will be calculated. This will be calculated separately for steps taken with each leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in a publication will be shared.
Time Frame: Relevant IPD and supporting information will be available within one year from when data is published, and will be available in perpetuity.
Access Criteria: Relevant IPD and supporting information will be shared through an accessible server online. Our current plan is to use the NIH BRICS data depository.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT07356011/Prot_SAP_000.pdf